CLINICAL TRIAL: NCT05689255
Title: A Prospective Cohort Study of Translational Changes in Gut Microbiome and Metabolome in Patients With Gallstone Disease After Surgical and Endoscopic Interventions
Brief Title: Gut Microbiome and Metabolome in Patients With Gallstone Disease After Surgical and Endoscopic Interventions
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Changi General Hospital (Other)
Responsible Party: Principal Investigator, Tiing Leong Ang, Senior Consultant, Department of Gastroenterology and Hepatology, Changi General Hospital
Other Study IDs: GMM1
Record Dates: First submitted 2022-11-28; First posted 2023-01-19 (Actual); Last update posted 2023-01-19 (Actual); Status verified 2023-01

CONDITIONS: Gallstone Disease; Bile Duct Diseases
Keywords: microbiome; metabolome
MeSH Terms: conditions — Cholelithiasis; Bile Duct Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Stool, plasma, urine and saliva before and after cholecystectomy; and bile following ERCP and endoscopic sphincterotomy
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this longitudinal observational cohort study is to examine the changes in the composition and diversity of gut microbiome and systemic metabolome in patients with symptomatic gallbladder stones with or without concomitant common bile duct (CBD) stones who will be undergoing cholecystectomy with or without prior endoscopic sphincterotomy (ERCP-ES) and CBD stones extraction. The main questions it aims to answer are whether there are:

* differences in gut microbiome diversity and composition before and after cholecystectomy
* differences in systemic metabolome before and after cholecystectomy
* gut microbiome and systemic metabolome changes after cholecystectomy

Participants will be asked to provide stool, urine, plasma and saliva samples prior to and 1-6 months after cholecystectomy. For patients with concomitant CBD stones who undergo ERCP-ES before cholecystectomy, bile specimens will be collected from the bile duct during ERCP-ES as well as the gallbladder and/or during cholecystectomy.

DETAILED DESCRIPTION:
This is a longitudinal observational cohort study that will examine the changes in the composition and diversity of gut microbiome and systemic metabolome in patients with symptomatic gallbladder stones with or without concomitant CBD stones who will be undergoing cholecystectomy with or without prior ERCP-ES and CBD stones extraction. This is a single centre study involving the Department of Gastroenterology and Hepatology and the Department of General Surgery at Changi General Hospital, SingHealth, Singapore.

Patients with symptomatic gallstones with or without CBD stones being planned for cholecystectomy will be recruited from both inpatient and outpatient settings. Upon enrolment, baseline clinical characteristics will be recorded, and biospecimens (stool, urine, plasma and saliva) will be collected prior to cholecystectomy for subsequent gut microbiome and systemic metabolome analysis. For patients with concomitant CBD stones who undergo ERCP-ES before cholecystectomy, bile specimens will be collected from the bile duct during ERCP-ES as well as the gallbladder during cholecystectomy, for subsequent bile microbiome analysis. After cholecystectomy, during the scheduled clinic review at 1 to 6 months post-surgery, patients will be reviewed for symptoms of post cholecystectomy syndrome (PCS) or post cholecystectomy diarrhoea (PCD), and biospecimens (stool, urine, plasma and saliva) will again be collected for subsequent gut microbiome and systemic metabolome analysis.

ELIGIBILITY:
Inclusion Criteria:

* Aged 21 years to 80 years
* Diagnosis of symptomatic gallstone disease without or with concomitant bile duct stones based on prior diagnostic radiological imaging such as transabdominal ultrasound (US), computed tomography (CT), magnetic resonance imaging (MRI) or endoscopic ultrasound (EUS).
* Will be scheduled for cholecystectomy with or without concomitant ERCP-ES for treatment.
* Patient is willing to provide informed consent before enrolment in the study.

Exclusion Criteria:

* Subjects undergoing ERCP-ES with no intention for future cholecystectomy
* Use of antibiotics or probiotics within 1 month (exception: use of antibiotics within 48 hours of cholecystectomy or ERCP, as metagenomics will be able to sequence both dead and live bacteria, and marked compositional change is not expected within this time frame)
* Presence of malignancy diagnosed within the last 1 year
* Previous gastrectomy, appendicectomy, small bowel or large bowel surgery
* Inflammatory bowel disease
* Active gastrointestinal tract infections

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This single centre study at Changi General Hospital will enrol up to 65 patients aged 21 to 80 years with symptomatic gallstone disease and/ or bile duct stones who will be undergoing cholecystectomy with or without concomitant ERCP-ES as part of standard clinical treatment. There will not be stratification by demographics.
Sampling Method: Non-Probability Sample
Enrollment: 65 (Estimated)
Dates: Start 2022-12-23 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Gut microbiome profile using metagenomic shotgun sequencing | 1-6 months
  Fresh stool samples will be collected for microbial DNA extraction prior to and 1-6 months after cholecystectomy. Microbial DNA will be extracted from the stool samples and used for metagenomic shotgun sequencing.
Systemic metabolome profile using targeted and untargeted metabolomic analysis | 1-6 months
  Urine, plasma and saliva samples will be collected for metabolomic profiling prior to and 1-6 months after cholecystectomy.

SECONDARY OUTCOMES:
Bile microbiome profile using metagenomic shotgun sequencing | 1-6 months
  Bile samples will be collected for microbial DNA extraction ERCP and endoscopic sphincterotomy

CONTACTS AND LOCATIONS:
Overall Officials: Tiing Leong Ang, Principal Investigator — Changi General Hospital
Locations (1):
- Changi General Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Reid FD, Mercer PM, harrison M, Bates T. Cholecystectomy as a risk factor for colorectal cancer: a meta-analysis. Scand J Gastroenterol. 1996 Feb;31(2):160-9. doi: 10.3109/00365529609031981. PMID 8658039
- [Background] Di Ciaula A, Garruti G, Wang DQ, Portincasa P. Cholecystectomy and risk of metabolic syndrome. Eur J Intern Med. 2018 Jul;53:3-11. doi: 10.1016/j.ejim.2018.04.019. Epub 2018 Apr 26. PMID 29706426
- [Background] Chen Y, Wu S, Tian Y. Cholecystectomy as a risk factor of metabolic syndrome: from epidemiologic clues to biochemical mechanisms. Lab Invest. 2018 Jan;98(1):7-14. doi: 10.1038/labinvest.2017.95. Epub 2017 Sep 11. PMID 28892095
- [Background] Latenstein CSS, Alferink LJM, Darwish Murad S, Drenth JPH, van Laarhoven CJHM, de Reuver PR. The Association Between Cholecystectomy, Metabolic Syndrome, and Nonalcoholic Fatty Liver Disease: A Population-Based Study. Clin Transl Gastroenterol. 2020 Apr;11(4):e00170. doi: 10.14309/ctg.0000000000000170. PMID 32352682